CLINICAL TRIAL: NCT05957133
Title: Comparison of the Effect on Functionality of Multicomponent Training With and Without Action Observation in Older Adults.
Brief Title: Effect of Action Observation Training in Older Adults.
Acronym: OAMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USalamancaAO
Record Dates: First submitted 2023-07-11; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Aging; Exercise
Keywords: exercise; elderly; multicomponent exercise; Action Observation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective, controlled, single-blind study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blind masking with blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise group without action observation (MTG) (Active Comparator): The main part of the multicomponent exercise program integrates different exercise modalities: Aerobic, mobility, strength, balance and coordination exercises, playful activities or games are also included with some activities aimed at working on cognitive functions to reinforce the overall effects of the program, such as games with colors, numbers, letters, right-left laterality, memory, etc.
  The progression of the different models is as follows:
  E. Aerobic: Start with continuous work, then intervallic, and decrease rest times in intervallic work.
  E. Strength: Increase sets, repetitions and decrease rest time. Balance: start with static and evolve with blindfolds, perturbations, dynamic balance, etc.
  Coordination, and cognitive games will also become more complicated, with more complicated and faster decision making.
  Interventions: Procedure: Multicomponent exercise without action observation.
- Multicomponent exercise group associated to action observation (AOG) (Experimental): It is the same intervention as the other group with the addition of the observation of actions thanks to the fact that the physiotherapist carries out the exercises with them at all times.
  The main part of the multicomponent exercise program integrates different exercise modalities: Aerobic, mobility, strength, balance and coordination exercises, playful activities or games are also included with some activities aimed at working on cognitive functions to reinforce the overall effects of the program, such as games with colors, numbers, letters, right-left laterality, memory, etc.
  The progression of the exercises will be the same as in the other group.
  Interventions: Procedure: Multicomponent exercise associated with action observation

INTERVENTIONS:
Procedure: Multicomponent exercise without action observation. — Different exercise modalities are integrated: Aerobic, mobility, strength, balance and coordination exercises.
  Arms: Multicomponent exercise group without action observation (MTG)
Procedure: Multicomponent exercise associated with action observation — Different exercise modalities are integrated: aerobic, mobility, strength, balance and coordination exercises carried out at all times by the physiotherapist and observed by the participants.
  Arms: Multicomponent exercise group associated to action observation (AOG)

SUMMARY:
Randomised clinical trial involving 58 independent subjects of both sexes who attended the Geriatric Revitalisation Programme run jointly by the University of Salamanca and the Salamanca City Council. At the beginning and at the end of the programme, data were collected on participants' balance, fall risk and other parameters, using anthropometric tests (weight, % body fat and body mass index (BMI)), and physical performance tests (grip strength, the Short Physical Performance Battery, TUG and the stair step test). Study participants performed three 50-minute sessions per week for a total of 35 weeks. The components of balance, gait, cardiovascular resistance, stability, upper and lower limb strength, flexibility and breathing exercises were worked on. In the OC group, the physiotherapist performed the entire session together with the participants, while in the other group, the physiotherapist simply ordered the exercises.

DETAILED DESCRIPTION:
Design: Randomised, controlled clinical trial with two parallel groups, in which adults over 65 years of age will be recruited. Study participants will be assigned to one of the two interventions. The study will have a duration of 35 weeks. There will be 2 evaluation visits, one initial, one final. During the intervention period there will be 3 weekly sessions of 50 minutes.

Scope: The study will be carried out in the Health Area of Salamanca, in collaboration with the Research, Teaching and Assistance Unit of the Faculty of Nursing and Physiotherapy of the University of Salamanca and the Department of Elderly People of the Salamanca City Council.

Interventions: 1) Multicomponent Exercise Group (GEM); 2) Multicomponent Exercise and Action Observation Group (GOA). The GEM and GOA sessions follow the same design, according to the recommendations of the American College of Sports Medicine (ACSM), the only difference being that in the GOA the physiotherapist will perform all the exercises with the participants.

Study population: Adults over 65 years of age from the city of Salamanca will be included, distributed in 2 groups in a 1:1 ratio. Randomisation will be performed using the Epidat 4.2 programme. The sample size was calculated using GRANMO Version 7. 12 April 2012.

The main study variables are: Functionality (Timed Up & Go test (TUG), chair stand test (CS), hand grip test (HG) and Short Physical Performance Battery (SPPB)), gait speed (GS). stair step test; and body composition (% body fat, body weight, body mass index (BMI)).

Population characteristics will be presented as mean and standard deviation for continuous variables and as frequency distribution for qualitative variables. Statistical analysis The effect of the intervention on the study variables if the variables are parametric Student's t-test will be used, and if they are non-parametric the Wilcoxon test will be used. An alpha risk of 0.05 is established as the limit of statistical significance. The statistical programme to be used will be SPSS, v.26.0.

The study will be carried out with the authorisation of the Ethics Committee for Research with Medicines (CEIm) of the Salamanca Health Area, and with the prior informed consent of the study subjects. Participants will be informed of the objectives of the project and of the risks and benefits of the tests and interventions to be performed. The study has been designed and subsequently evaluated in accordance with Law 14/2007 on Biomedical Research, the ethical principles of the Declaration of Helsinki of the World Medical Association on ethical principles for medical research on human beings, as well as the other ethical principles and legal regulations applicable according to the characteristics of the study.

ELIGIBILITY:
Inclusion Criteria:

* adults over 65 years of age.

Exclusion Criteria:

* Tumors
* Pacemakers
* Fibrillations
* Cardiac pathology or uncontrolled hypertension
* History of severe trauma/recent cervical surgery
* Uncontrolled systemic and inflammatory pathologies
* Congenital collagen compromise
* Presence of difficulties in performing the Initial Evaluation tests
* Language barriers
* Pending litigation or legal claim

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | thirty-five weeks
  Test to assess physical performance and degree of frailty consisting of 3 subtests: gait speed, balance, and lower limb strength. The maximum score is 12 points and a score ≤ 8 points indicates poor physical performance.

SECONDARY OUTCOMES:
Gait speed | thirty-five weeks
  It is considered a fast, safe and very reliable test, in a distance of 4 meters, values greater than 0.8 m/s are considered positive.
Timed Up and Go (TUG) | thirty-five weeks
  A predictive test for frailty and falls, where individuals are asked to get up from a standard chair, walk to a marker 3 m away, turn around, and sit down again. Times greater than 20 seconds are considered positive.
Grip strength test | thirty-five weeks
  Accurate measurement of hand grip strength requires the use of a calibrated hand dynamometer (Jamar Plus) under well-defined (standardised) test conditions. Force values below 16 kg are considered positive and indicate weakness.
Chair stand test | thirty-five weeks
  It can be used as an indicator of lower limb muscle strength. It measures the time it takes a patient to stand up five times from a seated position without using the arms. Times greater than 15 seconds are considered positive and indicate weakness.
Step-Up Box Test | thirty-five weeks
  Consists of climbing for two minutes on a 35 cm box as many times as possible. it trains the strength of the lower brain but also the cardiovascular resistance is assessed.
Body Mass Index (BMI) | thirty-five weeks
  It is a measure used to assess a person's body weight in relation to their height. It is calculated by dividing a person's weight in kilograms by their height in meters squared (BMI = kg/m²).
Body fat percentage | thirty-five weeks
  is total fat mass divided by total body mass, multiplied by 100. This is another obesity indicator like BMI.